CLINICAL TRIAL: NCT06240858
Title: Clinical Study of Self-gripping Mesh in Transabdominal Preperitoneal (TAPP) Versus Lichtenstein Hernia Repair
Brief Title: Clinical Study of Self-gripping Mesh in TAPP Versus Lichtenstein Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (2022) Annual Audit No. (175)
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Inguinal Hernia
Keywords: Self-gripping mesh; Laparoscopy; Herniorrhaphy
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAPP group (Experimental): The TAPP group underwent laparoscopic transperitoneal preperitoneal hernia repair.
  Interventions: Procedure: Laparoscopic transabdominal preperitoneal hernia repair.
- Lichtenstein group (Experimental): The Lichtenstein group underwent Lichtenstein hernia repair.
  Interventions: Procedure: Lichtenstein hernia repair.

INTERVENTIONS:
Procedure: Laparoscopic transabdominal preperitoneal hernia repair. — The TAPP group used self-gripping mesh for laparoscopic transperitoneal preperitoneal hernia repair.
  Arms: TAPP group
Procedure: Lichtenstein hernia repair. — The Lichtenstein group used self-gripping mesh for Lichtenstein hernia repair.
  Arms: Lichtenstein group

SUMMARY:
The goal of this prospective study is to compare the clinical efficacy of self-gripping mesh in laparoscopic transabdominal preperitoneal versus Lichtenstein hernia repair, in order to improve the outcome of inguinal hernia treatment. The main question it aims to answer is, in which procedure is the self-gripping mesh more effective.

Participants will be divided into the TAPP group and the Lichtenstein group by random number table method, the TAPP group underwent laparoscopic transperitoneal preperitoneal hernia repair, and the Lichtenstein group underwent Lichtenstein hernia repair, both groups used self-gripping meshes.

Researchers will compare the operation time, postoperative time out of bed, postoperative hospital stay, hospital costs and postoperative complications between the two groups to see the clinical efficacy of self-gripping mesh in laparoscopic transabdominal preperitoneal versus Lichtenstein hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years and older.
* Patients with a definite diagnosis of unilateral primary inguinal hernia.
* Patients and their families were informed about the study protocol and agreed to participate in the study.

Exclusion Criteria:

* Patients with femoral, recurrent, bilateral, incarcerated and strangulated hernias.
* Patients with previous history of lower abdominal surgery.
* Patients with contraindications to anaesthesia.
* Patients with contraindications to laparoscopic surgery.
* Failure to follow up patients as scheduled.
* Patients with abdominal infections.
* Those who cannot tolerate general anaesthesia surgery due to serious coagulation disorders, cardiopulmonary disorders, etc.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients aged 18 years and older were selected.
Enrollment: 130 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of moderate to severe pain at 3 and 6 months after surgery. | 3 and 6 months after surgery.
  Visual analogue scale (VAS) was used to score the postoperative pain at 3 and 6 months. The score ranges from 0 (no pain) to 10 (most severe pain).

SECONDARY OUTCOMES:
Incidence of recurrent inguinal hernia at 3 and 6 months after surgery. | 3 and 6 months after surgery.
  Recurrence of inguinal hernia after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
Data sharing with other researchers is not planned at this time due to patient privacy concerns.